CLINICAL TRIAL: NCT03188588
Title: Observance of Long Term Oxygen Therapy in Chronic Inspiratory Disease Patients
Acronym: ObsO2
Status: Completed | Type: Observational
Sponsor: SOS Oxygene Mediterranee (Industry)
Collaborators: CHU Arnaud de Villeneuve MONTPELLIER (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2016-A01244-47
Record Dates: First submitted 2017-06-12; First posted 2017-06-15 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2017-06

CONDITIONS: Chronic Respiratory Disease; Hypoxemia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Long-term oxygen therapy (LTOT) is the reference treatment for chronic respiratory failure. This treatment is based on the principle of oxygen supplementation via a source to correct hypoxemia in patients. At present, adherence to this treatment is difficult to evaluate (reporting by patients), but the results of the literature show poor LTOT compliance. It is therefore important to accurately measure the oxygen consumption by patients and to understand the factors explaining LTOT compliance. The ultimate aim is to improve our patient management to make them more observant in order to improve the therapeutic efficacy of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* chronic respiratory disease patients with chronic hypoxemia
* First prescribed long term oxygenotherapy

Exclusion Criteria:

* patients with NIV and CPAP
* vital pronostic < 3 months

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients are recruited from pneumologia unit of hospital and from private pneumologists
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
oxygen use | 6 month
  time of oxygen use

SECONDARY OUTCOMES:
respiratory disease severity based on GOLD standards | baseline
quality of life assessed by a questionnaire (VQ-11) | baseline, 3 month and 6 month
precarity score assessed by a questionnaire (EPICE) | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Bourdin, Professor, Principal Investigator — CHU Montpellier, France
Locations (1):
- CHU Arnaud de Villeneuve, Montpellier, France

IPD SHARING:
Plan to Share IPD: No